CLINICAL TRIAL: NCT01873001
Title: An Open-Label Drug-Drug Interaction Study to Assess the Effect of Abiraterone (JNJ-589485) on the Pharmacokinetics of Pioglitazone Following Administration of Abiraterone Acetate (JNJ-212082) and Pioglitazone HCl Tablets in Healthy Male Subjects
Brief Title: A Study to Assess the Effect of Abiraterone (JNJ-589485) on the Pharmacokinetics of Pioglitazone Following Administration of Abiraterone Acetate (JNJ-212082) and Pioglitazone HCl Tablets in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR101970; 212082PCR1011 (Other: Janssen Research & Development, LLC); 2013-001408-12 (EudraCT Number)
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; Drug-drug Interaction; Pharmacokinetics; Abiraterone; JNJ-589485; Abiraterone acetate; JNJ-212082; Pioglitazone HCl
MeSH Terms: interventions — Pioglitazone; Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abiraterone acetate + pioglitazone HCl (Experimental): Participants will receive 15 mg pioglitazone on Day 1 (Period 1). On Day 8 (Period 2), participants will receive 1000 mg abiraterone acetate followed by 15 mg of pioglitazone one hour later.
  Interventions: Drug: Pioglitazone HCl; Drug: Abiraterone acetate

INTERVENTIONS:
Drug: Pioglitazone HCl — 15 mg tablet administered by mouth on Day 1, and Day 8 1 hour after study drug administration
Drug: Abiraterone acetate — 1000 mg tablets administered by mouth on Day 8

SUMMARY:
The purpose of this study is to evaluate the effects of abiraterone on the pharmacokinetics (study of what the body does to a drug) of pioglitazone when coadministered with abiraterone acetate in healthy adult male participants.

DETAILED DESCRIPTION:
This is an open-label (identity of assigned study drug will be known) single-dose drug-drug interaction study to assess the effect of abiraterone on pioglitazone. Approximately 16 healthy adult male participants will be enrolled in this study. The study consists of a screening phase, an open-label treatment phase consisting of 2 single-dose treatment periods, end-of-study or withdrawal assessments done upon completion of the 72-hour pharmacokinetic sampling on Day 11 of Period 2 or upon withdrawal, and a follow-up visit 5 to 7 days after the last study procedure. The total study length is 32 days. Participants will receive pioglitazone alone on Day 1 (Period 1) of the study. On Day 8 (Period 2), participants will receive a single dose of abiraterone acetate followed by a single dose of pioglitazone one hour later. Successive pioglitazone administrations will be separated by a washout period of 7 days. Participants will be confined to the study center from Day -1 to Day 4 of Period 1 and from Day 7 to Day 11 of Period 2, at least 10 hours before each study drug administration until completion of the 72-hour blood sample collection for each period. A pharmacogenomic blood sample will be collected from all participants on Day -1. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Agrees to protocol-defined use of effective contraception for 1 week after receiving the last dose of study drug
* Agrees to not donate sperm during the study and for 1 week after receiving the last dose of study drug
* Body mass index between 18 and 30 kg/m2 and body weight not less than 50 kg
* Blood pressure between 90 and 140 mmHg systolic, and no higher than 90 mmHg diastolic
* A 12-lead electrocardiogram consistent with normal cardiac conduction and function
* Non-smoker
* Laboratory values within protocol -defined parameters

Exclusion Criteria:

* History of or current clinically significant medical illness
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or at admission to the study center as deemed appropriate by the investigator
* Presence of sexual dysfunction or any medical condition that would affect sexual function
* Clinically significant abnormal physical examination, vital signs, or 12-lead electrocardiogram
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements) before the first dose of the study drug is scheduled through study completion
* History of drug or alcohol abuse within 3 years before screening or positive test result(s) for alcohol and/or drugs of abuse at screening and Day -1 and at Day 7 of the treatment period
* Known allergy to the study drug or any of the excipients of the formulation
* History of stomach or intestinal surgery or resection that would potentially alter absorption or excretion of orally administered drugs (appendectomy and hernia repair will be allowed)
* Donated blood or blood products or had substantial loss of blood within 3 months before the first administration of study drug or intention to donate blood or blood products during the study
* Received an experimental drug or used an experimental medical device within 1 month or within a period less than 10 times the drug's half-life, whichever is longer, before the first dose of the study drug is scheduled
* Positive test for human immunodeficiency virus 1 and 2 antibodies, hepatitis B surface antigen, hepatitis B core antibody or hepatitis C antibodies
* Preplanned surgery or procedures that would interfere with the conduct of the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration of pioglitazone | Day 1 and Day 8 predose, and postdose at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h
Time to reach the maximum observed plasma concentration of pioglitazone | Day 1 and Day 8 predose, and postdose at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h
Area under the plasma concentration-time curve from time 0 to time of the last observed quantifiable concentration of pioglitazone | Day 1 and Day 8 predose, and postdose at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h
Area under the plasma concentration-time curve from time 0 to infinite time of pioglitazone | Day 1 and Day 8 predose, and postdose at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h
Percentage of area under the plasma concentration time curve obtained by extrapolation of pioglitazone | Day 1 and Day 8 predose, and postdose at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h
Elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve of pioglitazone | Day 1 and Day 8 predose, and postdose at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h
Time to last observed quantifiable plasma concentration of pioglitazone | Day 1 and Day 8 predose, and postdose at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h

SECONDARY OUTCOMES:
Maximum observed plasma concentration of abiraterone | Day 8 predose, and postdose at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h
Time to reach the maximum observed plasma concentration of abiraterone | Day 8 predose, and postdose at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h
Area under the plasma concentration-time curve from time 0 to time of the last observed quantifiable concentration of abiraterone | Day 8 predose, and postdose at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h
Area under the plasma concentration-time curve from time 0 to infinite time of abiraterone | Day 8 predose, and postdose at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h
Percentage of area under the plasma concentration-time curve obtained by extrapolation of abiraterone | Day 8 predose, and postdose at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h
Elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve of abiraterone | Day 8 predose, and postdose at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h
Time to last observed quantifiable plasma concentration of abiraterone | Day 8 predose, and postdose at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h
Apparent total plasma clearance of drug after extravascular administration of pioglitazone | Day 8 predose, and postdose at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h
Metabolite to parent drug ratio for maximum observed plasma concentration | Day 1 and Day 8 predose, and postdose at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h
Metabolite to parent drug ratio for area under the plasma concentration time curve from time 0 to time of the last observed quantifiable concentration | Day 1 and Day 8 predose, and postdose at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h
Metabolite to parent drug ratio for area under the plasma concentration time curve from time 0 to infinite time | Day 1 and Day 8 predose, and postdose at 30 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 36 h, 48 h, 72 h
Number of participants affected by adverse events by MedDRA system organ class (SOC) and Preferred term (PT) | Up to 30 days after the last dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium